CLINICAL TRIAL: NCT04532021
Title: Umbilical Cord and Maternal Blood Concentrations of Matrix Metalloproteinase 14, Neopterin, and Orosomucoid 1 in Pregnancy Complicated by Preterm Premature Rupture of the Membranes and Histological Chorioamnionitis
Brief Title: Matrix Metalloproteinase 14, Neopterin, and Orosomucoid 1 Levels in PPROM
Acronym: MMP-14&PPROM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH9
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Preterm Premature Rupture of Membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm premature rupture of membranes: Preterm premature rupture of membranes is the rupture of membranes during pregnancy before 37 weeks' gestation.
  Interventions: Diagnostic Test: matrix metalloproteinase 14, neopterin, and orosomucoid 1 measurements
- control group: Healthy subjects who had a normal pregnancy and outcomes without any fetal-neonatal complications will be accepted into the control group. Forty-four gestational age-matched healthy pregnant women who will be delivered at term will be included in the study as the control group.
  Interventions: Diagnostic Test: matrix metalloproteinase 14, neopterin, and orosomucoid 1 measurements

INTERVENTIONS:
Diagnostic Test: matrix metalloproteinase 14, neopterin, and orosomucoid 1 measurements — These three markers levels will be measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.

SUMMARY:
Introduction: To evaluate the maternal blood serum matrix metalloproteinase 14, neopterin, and orosomucoid 1 levels in pregnant women complicated by preterm premature rupture of membranes (PPROM) and to compare the results with healthy pregnancies. In addition, to determine whether maternal/umbilical cord blood concentrations of matrix metalloproteinase 14, neopterin, and orosomucoid 1 are of value in the diagnosis of histological chorioamnionitis in patients with preterm premature rupture of membranes (PPROM).

Methods: This cohort study will be included 44 pregnant women with PPROM and 44 gestational age-matched healthy subjects in 24-32 weeks of pregnancy. The blood for analysis will be firstly obtained in maternal blood on the day of diagnosis at the study group. Healthy subjects who have a normal pregnancy and outcomes without any fetal-neonatal complications will be accepted into the control group. Forty-four gestational age-matched healthy pregnant women who will be delivered at term will be included in the study as the control group. In the control group, the pregnant women will be taken the maternal blood at the admission day. The women in both groups will be observed until the delivery and perinatal data will be noted. Then, the blood for analysis will be secondly obtained in maternal blood during termination of the pregnancy (or spontaneous labor) at the study group. Lastly, the blood for analysis will be also obtained in umbilical cord blood at the study group. These three markers levels will be measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit. The placenta will be sent to histological examination in the study group. These three markers levels in women with PPROM will be compared to those of volunteer healthy pregnant women. In the study group, these three markers levels at maternal serum and cord serum will be evaluated for histological chorioamnionitis and maternal/neonatal outcomes.

DETAILED DESCRIPTION:
This observational case-control study will be conducted at the Department of Obstetrics and Gynecology, Cengiz Gokcek Public Hospital, Gaziantep, Turkey, between August 2020 and August 2021. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (reference no: 2020/212). The study strictly will be adhered to the principles of the Declaration of Helsinki. All subjects will be included in the study gave oral and written informed consent. Membrane rupture before labor and before 37 weeks of gestation is referred to as preterm premature rupture of membranes (PPROM). Every woman in the study population will be undergone obstetric ultrasound examination and fetal-maternal assessment will be carried out. The blood for analysis will be firstly obtained in maternal blood on the day of diagnosis at the study group. Healthy subjects who had a normal pregnancy and outcomes without any fetal-neonatal complications will be accepted into the control group. Forty-four gestational age-matched healthy pregnant women who will be delivered at term will be included in the study as the control group. In the control group, the pregnant women will be taken the maternal blood at the admission day. The women in both groups will be observed until the delivery and perinatal data will be noted. All The participants with PPROM will be also hospitalized. Then, the protocols for pregnant women with PPROM in our hospital are as follows: All patients with PPROM are hospitalized and expectant protocol is applied. After hospitalization until the delivery of baby, all pregnant women with PPROM receive prophylactic antibiotics for 1 week and betamethasone injection. The non-stress test and fetal movement determined by the mother are used for the detection of fetal well-being. The signs for clinical chorioamnionitis such as uterine tenderness, fever, purulent discharges from the cervical canal and inflammatory markers like white blood cell count (WBC) and C-reactive protein (CRP) levels are monitored carefully during the hospitalization. After a latency period, PPROM pregnancy will gone to spontaneous delivery or will be applied termination procedure. In the study group, the placenta will be stained with hematoxylin-eosin and will be examined under a light microscope for histological signs of neutrophil infiltration and chorioamnionitis. Then, this study will be determined maternal serum matrix metalloproteinase 14, neopterin, and orosomucoid 1 levels in women with PPROM(n=44) compared to those of volunteer healthy pregnant women (n=44). Then, these three markers levels at maternal serum and cord serum will be evaluated for histological chorioamnionitis and maternal/neonatal outcomes in the study group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women complicated with PPROM
* Healthy pregnant women who will be delivered at term
* Singleton pregnancy

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, renal disease and )
2. women who have dyed their hair in the last 9 months
3. history of using any medication
4. presence of gestational hypertension or gestational diabetes
5. drug user
6. patients who had fetal congenital abnormalities or genetic syndromes
7. multiple-gestation pregnancies
8. intrauterine fetal death
9. women who had any other infection or fever
10. fetal distress at admission
11. cord prolapse
12. active labor
13. antenatal bleeding
14. cervical or uterine anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — PPROM Preterm premature rupture of membranes (PPROM) is defined as the prelabor rupture of membranes before 37 weeks' gestation. Preterm PROM complicates about 1% of deliveries overall.
Study Population: The investigators consecutively will be recruited 44 subjects with PPROM, and 44 healthy pregnancies will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
MMP-14 levels in PPROM | 1 week
  The primary outcome in these analyses will compare maternal serum matrix metalloproteinase 14, neopterin, and orosomucoid 1 concentrations in PPROM group and control group.
neopterin levels in PPROM | 1 week
  The other primary outcome in these analyses will compare maternal serum neopterin concentrations in PPROM group and control group.
orosomucoid 1 levels in PPROM | 1 week
  The primary outcome in these analyses will compare maternal serum orosomucoid 1 concentrations in PPROM group and control group.

SECONDARY OUTCOMES:
markers levels for histological chorioamnionitis in PPROM | 1 week
  The secondary result in these analyzes will compare whether there is a difference at the levels of these three markers in maternal serum and cord serum for the presence of histological chorioamnionitis in the study group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Children's Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ekstrom B, Berggard I. Human alpha1-microglobulin. Purification procedure, chemical and physiochemical properties. J Biol Chem. 1977 Nov 25;252(22):8048-57. No abstract available. PMID 72071
- [Result] Nergiz Avcioglu S, Demircan Sezer S, Kucuk M, Zafer E, Yuksel H, Akcan B, Turgut O. Maternal serum concentrations of s-Endoglin and IL-6 in pregnancy complicated by preterm premature membrane rupture. J Matern Fetal Neonatal Med. 2016;29(12):1957-62. doi: 10.3109/14767058.2015.1070137. Epub 2015 Aug 13. PMID 26169712
- [Result] Hawinkels LJ, Kuiper P, Wiercinska E, Verspaget HW, Liu Z, Pardali E, Sier CF, ten Dijke P. Matrix metalloproteinase-14 (MT1-MMP)-mediated endoglin shedding inhibits tumor angiogenesis. Cancer Res. 2010 May 15;70(10):4141-50. doi: 10.1158/0008-5472.CAN-09-4466. Epub 2010 Apr 27. PMID 20424116
- [Result] Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 188: Prelabor Rupture of Membranes. Obstet Gynecol. 2018 Jan;131(1):e1-e14. doi: 10.1097/AOG.0000000000002455. PMID 29266075
- See also: a Citation — https://www.degruyter.com/view/journals/pteridines/14/1/article-p1.xml

DOCUMENTS (1):
  • Study Protocol (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT04532021/Prot_000.pdf